CLINICAL TRIAL: NCT04044703
Title: The VANcomycin Cohort Study - Assessing Precise Dosing and Prompt Drug Monitoring to Improve Attainment of Target Concentrations (Part 1)
Brief Title: Improving Dosing of Vancomycin in Young Infants With Infections
Acronym: VANCAPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Royal Hospital For Women (Other); University of Otago (Other); Sydney Children's Hospitals Network (Other); Monash Health (Other)
Responsible Party: Principal Investigator, Amanda Wilkins, Paediatric trainee, Murdoch Childrens Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC2019.059
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Infection; Bacteremia
MeSH Terms: conditions — Sepsis; Infections; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Model-based vancomycin dosing (Experimental): Participants will receive model-based intermittent intravenous vancomycin dosing as calculated by the dosing calculator available on a web application. Participants will then have routine therapeutic drug monitoring and linear dose adjustments.
  Interventions: Drug: Vancomycin - model-based dosing regimen

INTERVENTIONS:
Drug: Vancomycin - model-based dosing regimen — A dosing calculator based on a population pharmacokinetic model for vancomycin will be used to generate a participant's intermittent vancomycin dosing regimen. The participant's post-menstrual age, weight, creatinine and the target trough vancomycin level will be entered into the dosing calculator and the dose will be generated (intermittent infusion, dosing frequency will be from 1 to 4 times per day according to the corrected gestational age).

SUMMARY:
Current dosing regimens for vancomycin result in many young infants not reaching the target level of vancomycin in the blood at steady state (when the blood is in equilibrium at 24-48 hours).The purpose of this study is to assess an improved method of calculating the dose of vancomycin ('model-based dosing') in young infants with infections in order for them to achieve the target vancomycin level at steady state. A dosing calculator (which will be available through a web application) will be used for the dose calculation.

DETAILED DESCRIPTION:
Standard of care dosing of vancomycin in young infants is based on weight (eg. 15 mg/kg/dose). There is evidence that many young infants who are prescribed vancomycin using this calculation will not have enough vancomycin in the blood at steady state to treat an infection effectively. In this study a dosing calculator will be used to generate each participant's dose with the aim to improve the number of participant's who achieve the target vancomycin level (10 - 20 mg/L) at steady state. The dosing calculator is based on a pharmacokinetic/pharmacodynamic model of vancomycin which was built from prospective data. The participant's weight, post-menstrual age, creatinine and target vancomycin level will be entered into the dosing calculator (available on a web application), and the calculator will provide the dosing regimen for that participant. The participant will have the vancomycin level checked at 24-48 hours to assess if the target level has been achieved.

This study is 'part 1' of the study protocol (version 4.0) as approved under HREC reference number HREC/51942/RCHM-2019. This protocol also includes a second study, 'part 2', which will be registered with clinicaltrials.gov separately. Part 2 will assess the use of early drug monitoring and early dose adjustment to achieve the target vancomycin level in the blood at steady state. Part 1 of this protocol will be completed before part 2 begins recruitment. Part 1 and part 2 are two separate studies and the results of each part will not be compared to one another. However, each part will be compared to a retrospective control arm - infants from the VANC randomized controlled trial (NCT02210169) who received standard intermittent infusion of vancomycin dosing (as per British National Formulary for children. 15mg/kg/dose) and standard therapeutic drug monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0 - 90 days old
* Suspected infection requiring treatment with vancomycin for 48 hours or more (as determined by the clinical team)
* Post-Menstrual age (PMA) matched to PMA-group from retrospective control group

Exclusion Criteria:

* Infants with corrected gestational age of less than 25 weeks
* Infants weighing less than 500g
* Known allergy to any glycopeptide antibiotic
* Vancomycin administered within the previous 72 hours
* Infants receiving any form of extracorporeal life support
* Renal impairment
* Previously enrolled in the study

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
The proportion of young infants achieving target trough vancomycin concentrations (10 to 20 mg/L) at the first steady-state level when using a model-based dosing regimen | From first vancomycin dose (immediately after consent) to steady state level taken at 24-48 hours post-first-dose.

SECONDARY OUTCOMES:
The proportion of young infants with supra- (defined as >20mg/L) or sub- (defined as <10mg/L) therapeutic vancomycin concentrations at the first steady state level using a model-based dosing regimen (through a web application) | From first vancomycin dose (immediately after consent) to steady state level taken at 24-48 hours post-first-dose.
The proportion of young infants who are excluded from the study due to the model-based dosing regimen providing a total daily dose which exceeds 80 mg/kg/day despite a target trough concentration of 10 mg/L. | From consent to calculation of vancomycin dose (immediately after consent)
The frequency of drug-related adverse events (including infusion-related adverse events and nephrotoxicity). | From first vancomycin dose (immediately after consent) to completion of vancomycin therapy (as determined by clinical team, an average of 5 days)
The frequency of drug administration errors | From first vancomycin dose to completion of vancomycin therapy (as determined by clinical team, an average of 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wilkins, MBBS, Principal Investigator — Murdoch Childrens Research Institute
Locations (4):
- Australia (4):
  - Royal Hospital for Women, Sydney, New South Wales
  - Children's Hospital at Westmead, Sydney, New South Wales
  - Royal Children's Hospital Melbourne, Melbourne, Victoria
  - Monash Children's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No